CLINICAL TRIAL: NCT07004686
Title: Effect of MGRNOX-Guided General Anesthesia on Opioid Consumption in Patients:A Randomized Controlled Trial
Brief Title: Effect of MGRNOX-Guided General Anesthesia on Opioid Consumption in Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-024
Record Dates: First submitted 2025-05-18; First posted 2025-06-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGRNOX index-guided analgesia group (Experimental): After anesthesia induction, the remifentanil plasma target concentration was adjusted intraoperatively to maintain the MGRNOX index within 30-50,but mean arterial pressure and heart rate were additionally monitored and considered.
  Interventions: Device: MGRNOX index-guided analgesia
- Standard Clinical Care Group (Placebo Comparator): After anesthesia induction, the remifentanil plasma target concentration was adjusted intraoperatively based on mean arterial pressure and heart rate.
  Interventions: Device: Standard Clinical Care

INTERVENTIONS:
Device: MGRNOX index-guided analgesia — After anesthesia induction, the remifentanil plasma target concentration was adjusted intraoperatively to maintain the MGRNOX index between 30 and 50,but MAP and HR also were considered .In case the MGRNOX index was below 30 for more than 1 minute, remifentanil target-controlled infusion levels were lowered in steps of 0.5 ng/ml , whereas in case of a value greater than 50 for more than 1 minute, remifentanil target-controlled infusion levels were increased in steps of 0.5 ng/ml.
  Arms: MGRNOX index-guided analgesia group
Device: Standard Clinical Care — After anesthesia induction, if hypertension (MAP > 100 mmHg) or tachycardia (heart rate > 90 bpm) persists for more than 2 minutes, remifentanil target-controlled infusion levels were increased in steps of 0.5 ng/ml.If there is no response to remifentanil or the MAP and HR exceed a certain threshold, then urapidil or esmolol will be administered.For hypotension (50 mmHg < MAP ≤ 60 mmHg) persisting for more than 2 minutes, remifentanil target-controlled infusion levels were lowered in steps of 0.5 ng/ml (lowest target plasma concentration that was allowed is 1 ng/ml), and 4μg of norepinephrine were given. If MAP ≤ 50 mmHg, remifentanil target-controlled infusion levels were lowered in steps of 0.5 ng/ml(lowest target plasma concentration that was allowed is 1 ng/ml), and 8μg of norepinephrine were given.
  Arms: Standard Clinical Care Group

SUMMARY:
1. Pain management is a crucial part of general anesthesia surgery. Nociception monitoring can help anesthesiologists better titrate the use of intraoperative analgesic drugs, especially the opioid.
2. Although a variety of nociception monitoring devices have been developed to date, there is not a specific monitoring indicator that serves as the "gold standard" to objectively guide analgesic management in general anesthesia.
3. The MGRNOX index, which is derived from electroencephalogram (EEG), is used to reflect the correlation between noxious stimuli and opioid analgesics in a state of general anesthesia by converting and quantifying the EEG signals collected by the instrument. However, no studies have so far verified the effect of the MGRNOX index-guided analgesic management of general anesthesia on the consumption of opioids in patients.
4. This study aims to explore the effect of MGRNOX index-guided general anesthesia on opioid consumption in patients undergoing laparoscopic cholecystectomy and the primary hypothesis of our study is that using the MGRNOX index to guide intraoperative pain management during general anesthesia can significantly reduce the consumption of remifentanil during the surgery.

DETAILED DESCRIPTION:
Pain management is a critical component of perioperative anesthesia. Traditionally, anesthesiologists adjust analgesic dosages based on intraoperative heart rate or blood pressure, relying heavily on personal clinical experience. This approach often leads to over- or under-administration of analgesics. Currently, opioids remain the primary analgesics used in general anesthesia. Excessive opioid doses can result in postoperative hyperalgesia, delayed recovery, respiratory and circulatory depression, and increased hepatic/renal burden. Conversely, insufficient opioid doses may lead to inadequate analgesia, intraoperative hemodynamic instability, postoperative pain, and agitation.

In recent years, various nociception monitoring devices (e.g., SPI, ANI, qNOX) have been developed to quantify intraoperative nociception, assisting anesthesiologists in optimizing analgesic administration to achieve precision and balanced anesthesia. Studies suggest that nociception-guided analgesia during general anesthesia surgery reduces opioid consumption, alleviates postoperative pain, and improves hemodynamic stability compared to traditional standardized management. However, due to the limitations of existing indices, no specific parameter has yet been established as a gold standard for objectively reflecting intraoperative nociception levels.

The MGRNOX index, a China-developed metric based on central nervous system monitoring, derives from processed and quantified electroencephalographic (EEG) signals under general anesthesia to reflect a patient's analgesic state. As clinical evidence for MGRNOX remains limited and its impact on intraoperative opioid usage remains unvalidated, the investigators designed this randomized controlled trial to investigate whether MGRNOX-guided general anesthesia reduces opioid consumption during laparoscopic cholecystectomies. Our primary hypothesis is that intraoperative MGRNOX-guided analgesia will significantly decrease remifentanil requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and < 65 years old；
* American Society of Anesthesiologists (ASA) class I-II；
* Scheduled to undergo elective laparoscopic cholecystectomy undergeneral anesthesia （without epidural anesthesia, local blocks, or inﬁltration）

Exclusion Criteria:

* Pregnancy or lactation period；
* BMI ≥35 kg/m² or <18.5 kg/m²；
* Anticipated difficult airway；
* Previous diagnosis of hypertension；
* History of drug or alcohol abuse within the past 6 months；
* Preoperative acute or chronic pain history (routine preoperative use of opioid or non-opioid analgesics), peripheral or central nervous system-related disorders；
* Definitively diagnosed psychiatric disorders or other neuropsychiatric conditions severely affecting cognitive judgment, history of psychotropic medication use；
* Allergy or intolerance to anesthetic agents；
* Baseline mean arterial pressure (MAP) <60 mmHg or >120 mmHg; baseline heart rate (HR) <45 bpm or >90 bpm (Baseline values defined as first measurement taken in the ward after admission)；
* History of severe underlying diseases (untreated or ongoing peripheral/central cardiovascular diseases, severe hepatic disorders with elevated bilirubin/INR or hypoalbuminemia, severe renal diseases with elevated creatinine, severe pulmonary diseases potentially causing acute respiratory failure or persistent dyspnea)；
* Implanted pacemaker, chronic arrhythmia, preoperative use of prescribed anticholinergics, α2-adrenergic agonists, beta-1 adrenergic antagonists, or antiarrhythmic medications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
opioids | From the beginning of anesthesia induction until surgical procedure end（time of final wound closure）,assessed during surgery.
  Intraoperative remifentanil consumption, the dose unit is expressed as μg/kg/min.

SECONDARY OUTCOMES:
pain score | One hour after extubation
  The numerical rating scale (NRS，11-point scale, with 0 indicating no pain and 10 indicating the most severe pain) after extubation was evaluated every 15 minutes
Incidence of unexpected events | From the beginning of anesthesia induction until surgical procedure end（time of final wound closure）,assessed during surgery.
  severe hypotension：MAP<50mmHg，severe hypertension：MAP>120mmHg，tachycardia：HR>120beats/min，bradycardia：HR<40 beats/min，hypoxemia：SpO2≤92%，intraoperative awareness：Patients under general anesthesia showed a conscious state during the operation and could recall the surgery-related events that occurred during the operation postoperatively
incidence of complications | during PACU（at least 1 hour)
  postoperative complications during PACU：Nausea and vomiting，agitation，delirium
the consumption of sedative drug | From the beginning of anesthesia induction until 5 minutes before the end of the surgery.
  Intraoperative propofol consumption, the dose unit is expressed as mg/kg/h
the consumption of vasoactive drug | From the beginning of anesthesia induction until surgical procedure end（time of final wound closure）,assessed during surgery.
  Intraoperative vasoactive drugs consumption，involved drug type and dosage

CONTACTS AND LOCATIONS:
Overall Officials: Tao Luo, MD,PHD, Principal Investigator — Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Egan TD. Are opioids indispensable for general anaesthesia? Br J Anaesth. 2019 Jun;122(6):e127-e135. doi: 10.1016/j.bja.2019.02.018. Epub 2019 Mar 28. PMID 31104756
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Background] Kutlu Yalcin E, Araujo-Duran J, Turan A. Emerging drugs for the treatment of postsurgical pain. Expert Opin Emerg Drugs. 2021 Dec;26(4):371-384. doi: 10.1080/14728214.2021.2009799. Epub 2021 Nov 28. PMID 34842026
- [Background] Bergmann I, Gohner A, Crozier TA, Hesjedal B, Wiese CH, Popov AF, Bauer M, Hinz JM. Surgical pleth index-guided remifentanil administration reduces remifentanil and propofol consumption and shortens recovery times in outpatient anaesthesia. Br J Anaesth. 2013 Apr;110(4):622-8. doi: 10.1093/bja/aes426. Epub 2012 Dec 5. PMID 23220856
- [Background] Upton HD, Ludbrook GL, Wing A, Sleigh JW. Intraoperative "Analgesia Nociception Index"-Guided Fentanyl Administration During Sevoflurane Anesthesia in Lumbar Discectomy and Laminectomy: A Randomized Clinical Trial. Anesth Analg. 2017 Jul;125(1):81-90. doi: 10.1213/ANE.0000000000001984. PMID 28598927
- [Background] Jiang Y, Ding JM, Hao XX, Fang PP, Liu XS. EEG-derived pain threshold index-guided versus standard care during propofol-remifentanil anesthesia: A randomized controlled trial. Heliyon. 2023 Aug 1;9(8):e18604. doi: 10.1016/j.heliyon.2023.e18604. eCollection 2023 Aug. PMID 37593599
- [Background] Meijer F, Honing M, Roor T, Toet S, Calis P, Olofsen E, Martini C, van Velzen M, Aarts L, Niesters M, Boon M, Dahan A. Reduced postoperative pain using Nociception Level-guided fentanyl dosing during sevoflurane anaesthesia: a randomised controlled trial. Br J Anaesth. 2020 Dec;125(6):1070-1078. doi: 10.1016/j.bja.2020.07.057. Epub 2020 Sep 17. PMID 32950246
- [Background] Ma D, Ma J, Chen H, Mu D, Kong H, Yu L. Nociception monitors vs. standard practice for titration of opioid administration in general anesthesia: A meta-analysis of randomized controlled trials. Front Med (Lausanne). 2022 Aug 25;9:963185. doi: 10.3389/fmed.2022.963185. eCollection 2022. PMID 36091708
- [Background] Funcke S, Pinnschmidt HO, Brinkmann C, Wesseler S, Beyer B, Fischer M, Nitzschke R. Nociception level-guided opioid administration in radical retropubic prostatectomy: a randomised controlled trial. Br J Anaesth. 2021 Feb;126(2):516-524. doi: 10.1016/j.bja.2020.09.051. Epub 2020 Nov 20. PMID 33228979
- [Background] Renaud-Roy E, Morisson L, Brulotte V, Idrissi M, Godin N, Fortier LP, Verdonck O, Choiniere M, Richebe P. Effect of combined intraoperative use of the Nociception Level (NOL) and bispectral (BIS) indexes on desflurane administration. Anaesth Crit Care Pain Med. 2022 Jun;41(3):101081. doi: 10.1016/j.accpm.2022.101081. Epub 2022 Apr 25. PMID 35472586
- [Background] Coeckelenbergh S, Sessler DI, Doria S, Patricio D, Jaubert L, Huybrechts I, Stefanidis C, Kapessidou P, Tuna T, Engelman E, Barvais L, Perrin L. Nociception level index-guided antinociception versus routine care during remifentanil-propofol anaesthesia for moderate-to-high risk cardiovascular surgery: A randomized trial. Eur J Anaesthesiol. 2023 Oct 1;40(10):790-793. doi: 10.1097/EJA.0000000000001892. Epub 2023 Jul 26. No abstract available. PMID 37497778
- [Background] Meijer FS, Niesters M, van Velzen M, Martini CH, Olofsen E, Edry R, Sessler DI, van Dorp ELA, Dahan A, Boon M. Does nociception monitor-guided anesthesia affect opioid consumption? A systematic review of randomized controlled trials. J Clin Monit Comput. 2020 Aug;34(4):629-641. doi: 10.1007/s10877-019-00362-4. Epub 2019 Jul 20. PMID 31327102
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Background] Jiang Z, Xiao J, Wang X, Luo T. The effect-site concentration of remifentanil blunting endotracheal intubation responses during anesthesia induction with etomidate: a dose-finding study. BMC Anesthesiol. 2023 Jun 28;23(1):225. doi: 10.1186/s12871-023-02165-2. PMID 37380959
- [Background] Bourgeois C, Oyaert L, Van de Velde M, Pogatzki-Zahn E, Freys SM, Sauter AR, Joshi GP, Dewinter G; PROSPECT working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Pain management after laparoscopic cholecystectomy: A systematic review and procedure-specific postoperative pain management (PROSPECT) recommendations. Eur J Anaesthesiol. 2024 Nov 1;41(11):841-855. doi: 10.1097/EJA.0000000000002047. Epub 2024 Sep 3. PMID 39129451
- [Result] Meijer FS, Martini CH, Broens S, Boon M, Niesters M, Aarts L, Olofsen E, van Velzen M, Dahan A. Nociception-guided versus Standard Care during Remifentanil-Propofol Anesthesia: A Randomized Controlled Trial. Anesthesiology. 2019 May;130(5):745-755. doi: 10.1097/ALN.0000000000002634. PMID 30829658